CLINICAL TRIAL: NCT03252756
Title: Effects of Cannabidiol in Alcohol Use Disorder
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Tilray (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17-01001
Record Dates: First submitted 2017-08-14; First posted 2017-08-17 (Actual); Results first posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Alcohol Use Disorder
Keywords: Cannabidiol; Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized proof-of-concept study
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo for 4 weeks, followed by phytocannabinoid cannabidiol (CBD) for 4 weeks (Experimental): 600mg/day Saline taken by mouth (PO) for 4 weeks, immediately followed by 1200mg saline/ day (PO) for an additional 4 weeks (8 total weeks).
  Interventions: Other: Placebo
- CBD for 8 weeks (Experimental): 600mg CBD/day (PO) for 4 weeks, immediately followed by 1200mg CBD/day (PO) for an additional 4 weeks (8 total weeks).
  Interventions: Drug: Phytocannabinoid cannabidiol (CBD)

INTERVENTIONS:
Other: Placebo — Saline taken by mouth (PO)
  Arms: Placebo for 4 weeks, followed by phytocannabinoid cannabidiol (CBD) for 4 weeks
Drug: Phytocannabinoid cannabidiol (CBD) — CBD taken by mouth (PO)
  Arms: CBD for 8 weeks

SUMMARY:
The goal of the proposed project is to begin rigorous study of the clinically relevant effects of non-psychoactive phytocannabinoid cannabidiol (CBD) in patients with severe alcohol use disorder (AUD). This double-blind, randomized proof-of-concept study (n = 40) is designed to assess feasibility and contrast effects of extended (8 weeks) treatment with CBD to those of placebo in AUD patients. Participants with AUD will be randomized to receive either placebo or 600mg CBD/day (PO) for 4 weeks, immediately followed by 1200mg CBD/day (PO) for an additional 4 weeks (8 total weeks). These doses were chosen to reproduce serum CBD levels reported to reduce alcohol-seeking behavior in animal studies. Measures will include circulating levels of CBD, safety measures (THC serum levels, adverse events, cognitive and motoric function), and physiological and psychological domains relevant to AUD (including self-reported craving, depression, and anxiety, and responses to personalized scripts designed to elicit stress- and cue-induced craving and anxiety). Assessments will be conducted following 1 day, 1 week, and 4 weeks of treatment with each dose of CBD vs. placebo, and 1 and 4 weeks after the cessation of treatment. Drinking outcomes across 8 weeks of treatment and 4 weeks of follow-up will also be assessed as an exploratory outcome.

DETAILED DESCRIPTION:
There is increasing recognition of the roles of the endocannabinoid system in neurobiological processes and behavioral domains relevant to addiction. The non-psychoactive phytocannabinoid cannabidiol (CBD) has attracted considerable attention due to its lack of abuse potential, its excellent safety profile, its unique and complex pharmacology, and evidence that it affects anxiety and stress response in animal models and humans. There is a growing body of preclinical data demonstrating that CBD produces marked and persisting decreases in alcohol self-administration and preference for alcohol, and alcohol-, cue- and stress-induced reinstatement of alcohol-seeking behavior, yet there are few studies of the effects of CBD in humans with addictive disorders, and none in alcohol dependent patients.

ELIGIBILITY:
Inclusion Criteria:

* Males and females age 18-65
* DSM-5 diagnosis of moderate or severe AUD
* Able to provide voluntary informed consent
* At least 8 heavy drinking days (4 or more drinks for a woman, 5 or more drinks for a man) in the 30 days prior to screen
* If of childbearing potential (male or female), are willing to use approved form of contraception from screening for duration of the trial
* Able to provide at least two locators
* Endorse desire to cut down or stop drinking
* Agrees to abstain from all other cannabinoid use for duration of the study

Exclusion Criteria:

* Current alcohol withdrawal (CIWA-Ar score >7)
* Exclusionary medical conditions (e.g. current severe alcohol withdrawal requiring medical hospitalization, significantly impaired liver function)
* DSM-5 diagnosis of schizophrenia, schizoaffective disorder, bipolar disorder
* High risk of adverse emotional or behavioral reaction based on investigator's clinical evaluation (e.g., evidence of serious personality disorder, antisocial behavior, serious current stressors, lack of meaningful social support)
* Current significant suicidality (assessed using the C-SSRS), any suicidal behavior in the past 12 months, or any history of serious suicide attempts requiring hospitalization, or current significant homicidality
* History of severe Traumatic Brain Injury (LOC > 24 hours)
* DSM-5 diagnosis of current mild cannabis use disorder and/or moderate or severe substance use disorder for a substance other than alcohol or nicotine
* Significant laboratory abnormalities, including significantly impaired liver function, serious abnormalities of complete blood count or metabolic panel
* Active legal problems likely to result in incarceration within 12 weeks of treatment initiation
* Pregnancy or lactation
* Current use of exclusionary medications, including cannabinoids; treatments for addictions including alcohol; moderate to strong inhibitors of CYP3A4 or CYP2C19; medications metabolized primarily by CYP3A4, CYP3A5, or CYP3A7; and medications with a narrow therapeutic index which are substrates of UGT1A9, UGT2B7, CYP2C8, CYP2C9, CYP2C19, CYP1A2, or CYP2B6.
* Allergy to any ingredient of the study compound.
* Current treatment for AUD, with exception of AA/12-step treatment
* No inpatient psychiatric treatment in the last 12 months, with the exception of detox and extended Emergency Department stays
* A positive urine drug screen for THC, cocaine and/or opioids at screen

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2022-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bogenschutz, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal with have access to the data. To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Groups:
- 600mg Saline/Day for 4 Weeks, Then 1200mg Saline/Day for 4 Weeks: 600mg Saline/ day (PO) for 4 weeks, immediately followed by 1200mg Saline/ day (PO) for an additional 4 weeks (8 total weeks).
- 600mg CBD/Day for 4 Weeks, Then 1200mg CBD/Day for 4 Weeks: 600mg CBD/day for 4 weeks, immediately followed by 1200mg CBD/day for an additional 4 weeks (8 total weeks).
Period: Overall Study
Arm/Group | 600mg Saline/Day for 4 Weeks, Then 1200mg Saline/Day for 4 Weeks | 600mg CBD/Day for 4 Weeks, Then 1200mg CBD/Day for 4 Weeks
Started | 13 | 14
Completed | 10 | 8
Not Completed | 3 | 6
Not completed — Protocol Violation | 2 | 4
Not completed — COVID-19 Pandemic | 1 | 1
Not completed — Study Drug Expiration | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- 600mg Saline/Day for 4 Weeks, Then 1200mg Saline/Day for 4 Weeks: 600mg Saline (PO) for 4 weeks, immediately followed by 1200mg Saline/ day (PO) for an additional 4 weeks (8 total weeks).
- Total: Total of all reporting groups
Arm/Group | 600mg Saline/Day for 4 Weeks, Then 1200mg Saline/Day for 4 Weeks | 600mg CBD/Day for 4 Weeks, Then 1200mg CBD/Day for 4 Weeks | Total
Number analyzed (Participants) | 10 | 8 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.1 (9.71) | 37.75 (12.89) | 41.83 (11.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 8 | 6 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 8 | 6 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 7 | 3 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 10 | 8 | 18

OUTCOME MEASURES:

1. Primary Outcome: Trough CBD Plasma Levels
Description: CBD "trough" plasma levels measured before dosing with CBD.
Time Frame: Baseline
Measure: Median (Standard Deviation); unit: CBD (ng/mL)
Groups:
- Placebo: 600mg Saline (PO) for 4 weeks, immediately followed by 1200mg Saline/ day (PO) for an additional 4 weeks (8 total weeks).
- Phytocannabinoid Cannabidiol (CBD): 600mg CBD/day for 4 weeks, immediately followed by 1200mg CBD/day for an additional 4 weeks (8 total weeks).
Arm/Group | Placebo | Phytocannabinoid Cannabidiol (CBD)
Number analyzed (Participants) | 12 | 12
CBD (ng/mL) | 0 (0) | 0.7 (2.41)

2. Primary Outcome: Trough CBD Plasma Levels
Description: CBD "trough" plasma levels measured before dosing with CBD.
Time Frame: Week 1
Measure: Median (Standard Deviation); unit: CBD (ng/mL)
Arm/Group | Placebo | Phytocannabinoid Cannabidiol (CBD)
Number analyzed (Participants) | 11 | 12
CBD (ng/mL) | 0 (0) | 22.79 (16.44)

3. Primary Outcome: Trough CBD Plasma Levels
Description: CBD "trough" plasma levels measured before dosing with CBD.
Time Frame: Week 4
Measure: Median (Standard Deviation); unit: CBD (ng/mL)
Arm/Group | Placebo | Phytocannabinoid Cannabidiol (CBD)
Number analyzed (Participants) | 8 | 9
CBD (ng/mL) | 0.94 (2.66) | 31.21 (20.91)

4. Primary Outcome: Trough CBD Plasma Levels
Description: CBD "trough" plasma levels measured before dosing with CBD.
Time Frame: Week 5
Measure: Median (Standard Deviation); unit: CBD (ng/mL)
Arm/Group | Placebo | Phytocannabinoid Cannabidiol (CBD)
Number analyzed (Participants) | 9 | 8
CBD (ng/mL) | 0 (0) | 74.54 (44.85)

5. Primary Outcome: Trough CBD Plasma Levels
Description: CBD "trough" plasma levels measured before dosing with CBD.
Time Frame: Week 8
Measure: Median (Standard Deviation); unit: CBD (ng/mL)
Arm/Group | Placebo | Phytocannabinoid Cannabidiol (CBD)
Number analyzed (Participants) | 8 | 6
CBD (ng/mL) | 0 (0) | 100.03 (45.13)

6. Primary Outcome: Trough CBD Plasma Levels
Description: CBD "trough" plasma levels measured before dosing with CBD.
Time Frame: Week 9
Measure: Median (Standard Deviation); unit: CBD (ng/mL)
Arm/Group | Placebo | Phytocannabinoid Cannabidiol (CBD)
Number analyzed (Participants) | 9 | 6
CBD (ng/mL) | 0 (0) | 22.71 (19.67)

7. Primary Outcome: Peak CBD Plasma Levels
Description: CBD "peak" plasma levels measured 45 minutes after dosing with CBD.
Time Frame: Baseline
Measure: Median (Standard Deviation); unit: CBD (ng/mL)
Arm/Group | Placebo | Phytocannabinoid Cannabidiol (CBD)
Number analyzed (Participants) | 12 | 12
CBD (ng/mL) | 0 (0) | 52.04 (68.78)

8. Primary Outcome: Peak CBD Plasma Levels
Description: CBD "peak" plasma levels measured 45 minutes after dosing with CBD.
Time Frame: Day 1
Measure: Median (Standard Deviation); unit: CBD (ng/mL)
Arm/Group | Placebo | Phytocannabinoid Cannabidiol (CBD)
Number analyzed (Participants) | 11 | 11
CBD (ng/mL) | 0.67 (2.22) | 104.45 (99.24)

9. Primary Outcome: Peak CBD Plasma Levels
Description: CBD "peak" plasma levels measured 45 minutes after dosing with CBD.
Time Frame: Week 1
Measure: Median (Standard Deviation); unit: CBD (ng/mL)
Arm/Group | Placebo | Phytocannabinoid Cannabidiol (CBD)
Number analyzed (Participants) | 10 | 12
CBD (ng/mL) | 0 (0) | 83.67 (67.34)

10. Primary Outcome: Peak CBD Plasma Levels
Description: CBD "peak" plasma levels measured 45 minutes after dosing with CBD.
Time Frame: Week 4
Measure: Median (Standard Deviation); unit: CBD (ng/mL)
Arm/Group | Placebo | Phytocannabinoid Cannabidiol (CBD)
Number analyzed (Participants) | 8 | 9
CBD (ng/mL) | 0.94 (2.65) | 211.83 (197.34)

11. Primary Outcome: Peak CBD Plasma Levels
Description: CBD "peak" plasma levels measured 45 minutes after dosing with CBD.
Time Frame: Week 4 + 1 Day
Measure: Median (Standard Deviation); unit: CBD (ng/mL)
Groups:
- Phytocannabinoid Cannabidiol (CBD): 600mg CBD/day (PO) for 4 weeks, immediately followed by 1200mg CBD/day (PO) for an additional 4 weeks (8 total weeks).
Arm/Group | Placebo | Phytocannabinoid Cannabidiol (CBD)
Number analyzed (Participants) | 9 | 8
CBD (ng/mL) | 66.17 (198.52) | 102.74 (117.59)

12. Primary Outcome: Peak CBD Plasma Levels
Description: CBD "peak" plasma levels measured 45 minutes after dosing with CBD.
Time Frame: Week 5
Measure: Median (Standard Deviation); unit: CBD (ng/mL)
Arm/Group | Placebo | Phytocannabinoid Cannabidiol (CBD)
Number analyzed (Participants) | 9 | 8
CBD (ng/mL) | 0 (0) | 178.91 (211.35)

13. Primary Outcome: Peak CBD Plasma Levels
Description: CBD "peak" plasma levels measured 45 minutes after dosing with CBD.
Time Frame: Week 8
Measure: Median (Standard Deviation); unit: CBD (ng/mL)
Arm/Group | Placebo | Phytocannabinoid Cannabidiol (CBD)
Number analyzed (Participants) | 7 | 6
CBD (ng/mL) | 0 (0) | 275.012 (236.42)

14. Secondary Outcome: Percentage of Heavy Drinking Days
Description: The percent of heavy drinking days will be assessed by Timeline Follow Back (TLFB) methodology over the previous week. The TLFB methodology allows participants to report the number of days in the past 7 days in which they drank heavily.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Placebo | Phytocannabinoid Cannabidiol (CBD)
Number analyzed (Participants) | 12 | 13
percentage of days | 58.6 (30.10) | 46.67 (28.32)

15. Secondary Outcome: Percent of Heavy Drinking Days
Description: as for outcome 14
Time Frame: Week 1
Measure: Median (Standard Deviation); unit: percentage of days
Arm/Group | Placebo | Phytocannabinoid Cannabidiol (CBD)
Number analyzed (Participants) | 12 | 13
percentage of days | 35.71 (34.73) | 32.97 (32.15)

16. Secondary Outcome: Percent of Heavy Drinking Days
Description: as for outcome 14
Time Frame: Week 2
Measure: Median (Standard Deviation); unit: percentage of days
Arm/Group | Placebo | Phytocannabinoid Cannabidiol (CBD)
Number analyzed (Participants) | 10 | 11
percentage of days | 37.14 (37.45) | 17.86 (22.38)

17. Secondary Outcome: Percent of Heavy Drinking Days
Description: as for outcome 14
Time Frame: Week 3
Measure: Median (Standard Deviation); unit: percentage of days
Arm/Group | Placebo | Phytocannabinoid Cannabidiol (CBD)
Number analyzed (Participants) | 10 | 11
percentage of days | 32.86 (37.53) | 16.88 (24.59)

18. Secondary Outcome: Percent of Heavy Drinking Days
Description: as for outcome 14
Time Frame: Week 4
Measure: Median (Standard Deviation); unit: percentage of days
Arm/Group | Placebo | Phytocannabinoid Cannabidiol (CBD)
Number analyzed (Participants) | 10 | 10
percentage of days | 41.43 (35.28) | 21.43 (23.57)

19. Secondary Outcome: Percent of Heavy Drinking Days
Description: as for outcome 14
Time Frame: Week 5
Measure: Median (Standard Deviation); unit: percentage of days
Arm/Group | Placebo | Phytocannabinoid Cannabidiol (CBD)
Number analyzed (Participants) | 10 | 9
percentage of days | 15.71 (24.70) | 20.63 (28.67)

20. Secondary Outcome: Percent of Heavy Drinking Days
Description: as for outcome 14
Time Frame: Week 6
Measure: Median (Standard Deviation); unit: percentage of days
Arm/Group | Placebo | Phytocannabinoid Cannabidiol (CBD)
Number analyzed (Participants) | 10 | 9
percentage of days | 18.57 (31.62) | 20.63 (21.56)

21. Secondary Outcome: Percent of Heavy Drinking Days
Description: as for outcome 14
Time Frame: Week 7
Measure: Median (Standard Deviation); unit: percentage of days
Arm/Group | Placebo | Phytocannabinoid Cannabidiol (CBD)
Number analyzed (Participants) | 10 | 9
percentage of days | 18.57 (31.62) | 23.81 (20.20)

22. Secondary Outcome: Percent of Heavy Drinking Days
Description: as for outcome 14
Time Frame: Week 8
Measure: Median (Standard Deviation); unit: percentage of days
Arm/Group | Placebo | Phytocannabinoid Cannabidiol (CBD)
Number analyzed (Participants) | 10 | 9
percentage of days | 18.57 (22.39) | 12.70 (15.06)

23. Secondary Outcome: Percent of Heavy Drinking Days
Description: as for outcome 14
Time Frame: Week 9
Measure: Median (Standard Deviation); unit: percentage of days
Arm/Group | Placebo | Phytocannabinoid Cannabidiol (CBD)
Number analyzed (Participants) | 10 | 9
percentage of days | 24.29 (36.92) | 15.87 (15.06)

24. Secondary Outcome: Number of Drinks Per Day
Description: The number of drinks per day will be assessed by Timeline Follow Back (TLFB) methodology over the previous week. The TLFB methodology allows participants to report the number of drinks per day over the last 7 days.
Time Frame: Baseline
Measure: Median (Standard Deviation); unit: Drinks per day
Arm/Group | Placebo | Phytocannabinoid Cannabidiol (CBD)
Number analyzed (Participants) | 12 | 13
Drinks per day | 5.38 (2.40) | 4.61 (2.17)

25. Secondary Outcome: Number of Drinks Per Day
Description: as for outcome 24
Time Frame: Week 1
Measure: Median (Standard Deviation); unit: drinks per day
Arm/Group | Placebo | Phytocannabinoid Cannabidiol (CBD)
Number analyzed (Participants) | 12 | 13
drinks per day | 3.23 (2.55) | 2.91 (2.28)

26. Secondary Outcome: Number of Drinks Per Day
Description: as for outcome 24
Time Frame: Week 2
Measure: Median (Standard Deviation); unit: drinks per day
Arm/Group | Placebo | Phytocannabinoid Cannabidiol (CBD)
Number analyzed (Participants) | 10 | 11
drinks per day | 4.36 (5.30) | 2.37 (2.03)

27. Secondary Outcome: Number of Drinks Per Day
Description: as for outcome 24
Time Frame: Week 3
Measure: Median (Standard Deviation); unit: drinks per day
Arm/Group | Placebo | Phytocannabinoid Cannabidiol (CBD)
Number analyzed (Participants) | 10 | 11
drinks per day | 3.28 (3.17) | 1.83 (1.77)

28. Secondary Outcome: Number of Drinks Per Day
Description: as for outcome 24
Time Frame: Week 4
Measure: Median (Standard Deviation); unit: drinks per day
Arm/Group | Placebo | Phytocannabinoid Cannabidiol (CBD)
Number analyzed (Participants) | 10 | 10
drinks per day | 4.49 (3.36) | 2.13 (2.00)

29. Secondary Outcome: Number of Drinks Per Day
Description: as for outcome 24
Time Frame: Week 5
Measure: Median (Standard Deviation); unit: drinks per day
Arm/Group | Placebo | Phytocannabinoid Cannabidiol (CBD)
Number analyzed (Participants) | 10 | 9
drinks per day | 1.66 (1.92) | 2.39 (2.14)

30. Secondary Outcome: Number of Drinks Per Day
Description: as for outcome 24
Time Frame: Week 6
Measure: Median (Standard Deviation); unit: drinks per day
Arm/Group | Placebo | Phytocannabinoid Cannabidiol (CBD)
Number analyzed (Participants) | 10 | 9
drinks per day | 1.82 (2.39) | 2.38 (1.94)

31. Secondary Outcome: Number of Drinks Per Day
Description: as for outcome 24
Time Frame: Week 7
Measure: Median (Standard Deviation); unit: drinks per day
Arm/Group | Placebo | Phytocannabinoid Cannabidiol (CBD)
Number analyzed (Participants) | 10 | 9
drinks per day | 1.82 (2.39) | 2.57 (1.95)

32. Secondary Outcome: Number of Drinks Per Day
Description: as for outcome 24
Time Frame: Week 8
Measure: Median (Standard Deviation); unit: drinks per day
Arm/Group | Placebo | Phytocannabinoid Cannabidiol (CBD)
Number analyzed (Participants) | 10 | 9
drinks per day | 2.26 (2.73) | 1.99 (1.60)

33. Secondary Outcome: Number of Drinks Per Day
Description: as for outcome 24
Time Frame: Week 9
Measure: Median (Standard Deviation); unit: drinks per day
Arm/Group | Placebo | Phytocannabinoid Cannabidiol (CBD)
Number analyzed (Participants) | 10 | 9
drinks per day | 3.17 (4.28) | 2.40 (2.32)

34. Secondary Outcome: Penn Alcohol Craving Scale (PACS) Score
Description: 5-item self-report measure of alcohol craving. Items are ranked on a Likert scale ranging from 0 (not at all) to 6 (severely). The total score is a sum of all the responses and ranges from 0 to 30. Higher scores indicate greater alcohol craving.
Time Frame: Baseline
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Phytocannabinoid Cannabidiol (CBD)
Number analyzed (Participants) | 11 | 13
score on a scale | 14.20 (4.58) | 17.77 (5.46)

35. Secondary Outcome: Penn Alcohol Craving Scale (PACS) Score
Description: as for outcome 34
Time Frame: Week 1
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Phytocannabinoid Cannabidiol (CBD)
Number analyzed (Participants) | 11 | 11
score on a scale | 13.45 (7.16) | 14.09 (7.69)

36. Secondary Outcome: Penn Alcohol Craving Scale (PACS) Score
Description: as for outcome 34
Time Frame: Week 4
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Phytocannabinoid Cannabidiol (CBD)
Number analyzed (Participants) | 9 | 9
score on a scale | 13.67 (6.98) | 10.33 (4.56)

37. Secondary Outcome: Penn Alcohol Craving Scale (PACS) Score
Description: as for outcome 34
Time Frame: Week 5
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Phytocannabinoid Cannabidiol (CBD)
Number analyzed (Participants) | 9 | 9
score on a scale | 11.78 (6.51) | 11.78 (6.08)

38. Secondary Outcome: Penn Alcohol Craving Scale (PACS) Score
Description: as for outcome 34
Time Frame: Week 8
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Phytocannabinoid Cannabidiol (CBD)
Number analyzed (Participants) | 9 | 9
score on a scale | 10.22 (5.87) | 11.56 (5.10)

39. Secondary Outcome: Penn Alcohol Craving Scale (PACS) Score
Description: as for outcome 34
Time Frame: Week 9
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Phytocannabinoid Cannabidiol (CBD)
Number analyzed (Participants) | 9 | 6
score on a scale | 8.22 (5.40) | 11.33 (3.72)

40. Secondary Outcome: Beck Anxiety Inventory (BAI) Score
Description: 21-item self-report measure of anxiety. Items are ranked on a Likert scale ranging from 0 (Not at all) to 3 (Severely). The total score is the sum of responses and ranges from 0 to 63, where higher scores indicate greater levels of anxiety. Scores are interpreted as follows: 0 - 21 = low anxiety; 22 - 35 = moderate anxiety; 36 and above = potentially concerning levels of anxiety.
Time Frame: Baseline
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Phytocannabinoid Cannabidiol (CBD)
Number analyzed (Participants) | 12 | 13
score on a scale | 6.92 (5.12) | 8 (7.40)

41. Secondary Outcome: Beck Anxiety Inventory (BAI) Score
Description: as for outcome 40
Time Frame: Week 1
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Phytocannabinoid Cannabidiol (CBD)
Number analyzed (Participants) | 10 | 12
score on a scale | 5.6 (7.14) | 8 (8.81)

42. Secondary Outcome: Beck Anxiety Inventory (BAI) Score
Description: as for outcome 40
Time Frame: Week 4
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Phytocannabinoid Cannabidiol (CBD)
Number analyzed (Participants) | 9 | 9
score on a scale | 3.33 (4.39) | 11.33 (8.59)

43. Secondary Outcome: Beck Anxiety Inventory (BAI) Score
Description: as for outcome 40
Time Frame: Week 5
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Phytocannabinoid Cannabidiol (CBD)
Number analyzed (Participants) | 10 | 7
score on a scale | 2.4 (4.48) | 6.57 (9)

44. Secondary Outcome: Beck Anxiety Inventory (BAI) Score
Description: as for outcome 40
Time Frame: Week 8
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Phytocannabinoid Cannabidiol (CBD)
Number analyzed (Participants) | 9 | 9
score on a scale | 4 (6.24) | 6.67 (8.60)

45. Secondary Outcome: Beck Anxiety Inventory (BAI) Score
Description: as for outcome 40
Time Frame: Week 9
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Phytocannabinoid Cannabidiol (CBD)
Number analyzed (Participants) | 9 | 8
score on a scale | 1.89 (2.80) | 6.125 (9.46)

46. Secondary Outcome: Beck Depression Inventory (BDI) Score
Description: 21-item self-report measure of depression. Items are ranked on a Likert scale ranging from 0 (Not at all) to 3 (Severely). The total score is the sum of responses and ranges from 0 to 63, where higher scores indicate greater levels of depression. Scores are interpreted as follows: 0 - 10 = normal ups and downs; 11-16 = mild mood disturbance; 17-20 = borderline clinical depression; 21-30 = moderate depression; 31-40 = severe depression; over 40 = extreme depression.
Time Frame: Baseline
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Phytocannabinoid Cannabidiol (CBD)
Number analyzed (Participants) | 12 | 13
score on a scale | 9.25 (7.19) | 9.92 (7.89)

47. Secondary Outcome: Beck Depression Inventory (BDI) Score
Description: as for outcome 46
Time Frame: Week 1
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Phytocannabinoid Cannabidiol (CBD)
Number analyzed (Participants) | 10 | 12
score on a scale | 7.2 (7.64) | 7.83 (6.39)

48. Secondary Outcome: Beck Depression Inventory (BDI) Score
Description: as for outcome 46
Time Frame: Week 4
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Phytocannabinoid Cannabidiol (CBD)
Number analyzed (Participants) | 10 | 9
score on a scale | 5.2 (7.67) | 9 (7.07)

49. Secondary Outcome: Beck Depression Inventory (BDI) Score
Description: as for outcome 46
Time Frame: Week 5
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Phytocannabinoid Cannabidiol (CBD)
Number analyzed (Participants) | 10 | 9
score on a scale | 5.1 (8.94) | 7.67 (6.89)

50. Secondary Outcome: Beck Depression Inventory (BDI) Score
Description: as for outcome 46
Time Frame: Week 8
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Phytocannabinoid Cannabidiol (CBD)
Number analyzed (Participants) | 9 | 9
score on a scale | 4.67 (6.10) | 7.67 (7.57)

51. Secondary Outcome: Beck Depression Inventory (BDI) Score
Description: as for outcome 46
Time Frame: Week 9
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Phytocannabinoid Cannabidiol (CBD)
Number analyzed (Participants) | 9 | 8
score on a scale | 3.90 (3.92) | 6.5 (6.93)

ADVERSE EVENTS:
Time Frame: 12 Weeks
Description: Study clinicians monitored study participants for adverse events at every follow-up visit, and recorded information on a standardized adverse event form.
Arm/Group | Placebo | Phytocannabinoid Cannabidiol (CBD)
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 1/13
Other Adverse Events (participants affected / at risk) | 7/13 | 10/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=13) | Phytocannabinoid Cannabidiol (CBD) (N=13)
Hospitalization for Ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=13) | Phytocannabinoid Cannabidiol (CBD) (N=13)
Nausea (Gastrointestinal disorders) | 0 | 4
Runny Nose (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Muscle Pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Headache (Nervous system disorders) | 2 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Diarrhea (Gastrointestinal disorders) | 2 | 4
Fatigue (General disorders) | 0 | 2
Appetite Increase (Metabolism and nutrition disorders) | 0 | 2
Increased Bowl Movement (Gastrointestinal disorders) | 0 | 1
Body Ache (Musculoskeletal and connective tissue disorders) | 0 | 2
Gum Infection (Infections and infestations) | 0 | 1
Fever (Infections and infestations) | 0 | 2
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Irregular Heartbeat (Cardiac disorders) | 1 | 0
Light-Headedness (Nervous system disorders) | 2 | 0
Drowsy (Nervous system disorders) | 2 | 0
Suicidal Ideation (Psychiatric disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 3
Dry Mouth (Gastrointestinal disorders) | 2 | 2
Gum Problems (Gastrointestinal disorders) | 0 | 1
Stomach/Abdominal Discomfort (Gastrointestinal disorders) | 0 | 1
Taste Abnormality (Nervous system disorders) | 0 | 1
Cognitive Slowing (Psychiatric disorders) | 0 | 1
Increased Thirst (Metabolism and nutrition disorders) | 0 | 1
Queasiness (Gastrointestinal disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Euphoria (Psychiatric disorders) | 1 | 1
Perceptual Problems (Psychiatric disorders) | 1 | 2
Hair Problems (Skin and subcutaneous tissue disorders) | 0 | 1
Irritability (Psychiatric disorders) | 0 | 1
Feeling "High" (Psychiatric disorders) | 0 | 2
Perceptual Enhancement (Psychiatric disorders) | 0 | 1
Relaxed Breathing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tiredness/Fatigue (General disorders) | 1 | 0
Elevated Heptic Enzymes (Hepatobiliary disorders) | 1 | 1
Vivid Dreaming (Psychiatric disorders) | 1 | 1
Increased Alcohol Craving (Psychiatric disorders) | 1 | 0
Concentration Difficulty (Psychiatric disorders) | 1 | 2
Heartburn / Acid Reflux (Gastrointestinal disorders) | 0 | 1
Memory Problems (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 2
Loose Stool (Gastrointestinal disorders) | 0 | 1
Upper Respiratory Infection (Infections and infestations) | 0 | 1
Drowsiness (General disorders) | 0 | 1
Confusion (Psychiatric disorders) | 0 | 1
Rash / Skin Irritation (Skin and subcutaneous tissue disorders) | 0 | 1
Flu (Infections and infestations) | 0 | 1
Pink Eye (Eye disorders) | 0 | 1
Chills (General disorders) | 0 | 1
Vivid Dreams (Psychiatric disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-20): https://cdn.clinicaltrials.gov/large-docs/56/NCT03252756/Prot_SAP_000.pdf